CLINICAL TRIAL: NCT05604742
Title: Belimumab for Treatment of Chronic Graft-versus-Host Disease Following Allogeneic Hematopoietic Cell Transplantation
Brief Title: Belimumab for Treatment of cGVHD Following Allo-HCT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No patients eligible for inclusion
Sponsor: xuna (Other)
Responsible Party: Sponsor-Investigator, xuna, professor, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cGVHD202210310
Record Dates: First submitted 2022-10-30; First posted 2022-11-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: cGVHD
Keywords: cGVHD; Resistance; belimumab
MeSH Terms: interventions — belimumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-dose group of Belimumab (Experimental): Belimumab 1mg/kg com combined with conventional therapy
  Interventions: Drug: Belimumab (Benlysta)
- High-dose group of Belimumab (Experimental): Belimumab 4mg/kg com combined with conventional therapy
  Interventions: Drug: Belimumab (Benlysta)
- Control group (No Intervention): conventional therapy

INTERVENTIONS:
Drug: Belimumab (Benlysta) — Belimumab will be administered intravenously every 2 weeks for 3 cycles and then every 4 weeks for a total of 5 cycles
  Arms: High-dose group of Belimumab; Low-dose group of Belimumab

SUMMARY:
Given the role of B cells in the pathophysiology of chronic graft versus host disease (GvHD), the association between elevated BAFF levels post-transplant in abnormal B-cell homeostasis and chronic GvHD, and the efficacy of belimumab in the inhibition of soluble human B lymphocyte stimulator protein (BAFF) signaling, these proof-of-principle findings support the rational for use of belimumab as treatment of chronic GvHD.The investigators propose a pilot and feasibility study to assess the safety and tolerability, as well as preliminary efficacy, of belimumab a treatment of cGvHD following allogeneic hematopoietic cell transplantation (alloHCT). The investigators' central hypothesis is that belimumab will be well tolerated and have a favorable effect on chronic GvHD,and we explored therapeutic dosage of belimumab.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 65years old 2.Newly diagnosed, moderate or severe chronic GvHD according to the 2014 NIH Consensus Criteria, requiring systemic immunosuppression 3.Karnofsky performance status greater than or equal to 60% 4.History of prior alloHSCT; any donors, conditioning regimens and graft sources are allowed 5.Newly diagnosed moderate or severe chronic Graft versus Host Disease (GvHD) (according to the 2014 NIH Consensus Criteria, requiring systemic immunosuppression 6.History of prior allogeneic Hematopoietic Stem Cell Transplant (HSCT) (any donors, conditioning regimens and graft sources are allowed).

7.Stable doses of other immunosuppressive medications (e.g., calcineurin inhibitors, mycophenolate mofetil, rapamune, etc.) with no dose increase in the 2 weeks prior to study treatment initiation. Doses may be adjusted for trough levels.

8.Patients tested positive for autoantibodies (ANA titer ≥1:80) and high BAFF levels (plasma concentration ≥15ng/ml).

9.Laboratory parameters as defined below: Serum creatinine less than or equal to 2.0 x ULN AST and ALT less than or equal to 3 x ULN (less than or equal to 5 x ULN if unequivocal liver GvHD) Total bilirubin less than or equal to 3 x ULN 10.Ability to understand and willingness to sign a written informed consent fo

Exclusion Criteria:

1. Relapsed or progressive malignant disease (other than minimal residual disease)
2. History of other malignant diseases, including post-transplant lymphoproliferative disease
3. Rituximab or other anti-B cell-specific antibodies were used in the past 3 months.
4. Uncontrolled infections (including prior aspergillosis) not responsive to antibiotics, antiviral medicines, or antifungal medicines
5. Donor lymphocyte transfusion for donor chimeric relapse or loss.
6. Any other reason at the discretion of the investigators and documented in the medical record that may raise concerns about the subject safety or ability to participate on this study -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate of chronic GvHD after belimumab treatment | approximately 6 months
  cGVHD grade according NIH

SECONDARY OUTCOMES:
Duration of response rate of chronic GvHD after belimumab treatment | 12 months
  Duration of ORR chronic GvHD after belimumab treatment

OTHER OUTCOMES:
Safety and tolerability of belimumab as treatment of chronic GvHD | approximately 12 months
  Adverse events will be graded according to CTCAE v4.03.
Overall survival | 24 months
  Overall survival will be determined from date of belimumab initiation, with death from any cause as the event of interest, and censoring at last follow up date for those with incomplete observations.
  Overall survival will be determined from date of belimumab initiation, with death from any cause as the event of interest, and censoring at last follow up date for those with incomplete observations.
  Overall survival will be determined from date of belimumab initiation, with death from any cause as the event of interest, and censoring at last follow up date for those with incomplete observations.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Nanfang Hospital, Southern Medical University,, Guanzhou, China

IPD SHARING:
Plan to Share IPD: No